CLINICAL TRIAL: NCT05388032
Title: A Mechanistic Trial of Dietary Sodium Reduction on Vascular Structure and Function
Brief Title: Sodium Lowering Vascular Effects Trial
Acronym: SOLVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Katherine T Mills, Associate Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01HL155559 (NIH)
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Endothelial Dysfunction; Vascular Stiffness; Left Ventricular Hypertrophy; Left Ventricular Dysfunction
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1 into the dietitian-led behavioral intervention and usual diet.
Who Masked: Outcomes Assessor
Masking Description: Clinical and laboratory staff members who assess the study outcomes will be blinded to participant intervention assignment. Study participants, investigators, and study staff members who conduct the intervention cannot be blinded to intervention assignment because this is a dietary behavioral intervention trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium reduction intervention (Experimental): The sodium reduction intervention is a dietician-led behavioral intervention consisting of two phases, first a 3-month intensive intervention phase, followed by a 9-month maintenance phase. The overall goal of the intervention is to reduce sodium intake to <2,300 mg per day based on the most recent guideline from the National Academies of Medicine. Both phases will include individual and group behavioral modification counseling designed to facilitate a reduction in dietary sodium intake.
  Interventions: Behavioral: Sodium Reduction Intervention
- Usual Diet (No Intervention): Participants randomized to the usual diet group will receive standard care from their providers with no study intervention.

INTERVENTIONS:
Behavioral: Sodium Reduction Intervention — The sodium reduction intervention is a dietician-led behavioral intervention consisting of two phases, first a 3-month intensive intervention phase, followed by a 9-month maintenance phase. The overall goal of the intervention is to reduce sodium intake to <2,300 mg per day based on the most recent guideline from the National Academies of Medicine. Both phases will include individual and group behavioral modification counseling designed to facilitate a reduction in dietary sodium intake.
  Arms: sodium reduction intervention

SUMMARY:
The proposed mechanistic trial will test the effect of dietary sodium reduction on cardiac and vascular structure and function in those with elevated blood pressure or hypertension. Findings from this study will fill the knowledge gap on the underlying mechanisms of dietary sodium intake on cardiovascular disease risk in addition to blood pressure and could provide further evidence on sodium reduction for the prevention of cardiovascular disease.

DETAILED DESCRIPTION:
High dietary sodium intake increases risk of cardiovascular disease (CVD) independent of established risk factors, including blood pressure (BP). Non-BP mediated mechanisms underlying the increased risk of CVD associated with dietary sodium intake are not well understood, but observational studies suggest direct target organ damage in the heart and vasculature might play an important role. Little evidence exists from randomized controlled trials (RCTs) on target organ effects of dietary sodium reduction, and the National Academy of Medicine has recommended future research to "test the effects of different sodium intake levels on endothelial and vascular function" in order to "to better characterize the relationship between sodium intake and chronic disease". The overall objective of the proposed mechanistic trial is to test the effect of dietary sodium reduction on cardiac and vascular structure and function. Specifically, the proposed trial will test whether dietary sodium reduction (targeting a dietary sodium intake of <2,300 mg/day) will improve left ventricular mass index (LVMI), left ventricular global longitudinal strain (LVGLS), carotid-femoral pulse wave velocity (cfPWV), and flow-mediated dilation (FMD) compared to usual intake. Additionally, we will test whether this effect is independent from BP reduction. We will recruit 256 people with elevated BP or hypertension from the greater New Orleans area and randomly assign them to a dietitian-led behavioral intervention aimed at decreasing dietary sodium intake to <2,300 mg/day for 12 months or to a usual diet. Study outcomes, including cardiac magnetic resonance imaging (CMR)-determined LVMI and LVGLS, cfPWV, and FMD, will be measured at baseline, 6-month, and 12-month clinic visits using standardized protocols with stringent quality control. These outcomes are validated biomarkers for target organ damage and predict the risk of clinical CVD events. In primary analyses, the effect of sodium reduction on each subclinical CVD endpoint will be compared between the sodium reduction and usual diet groups according to the intention-to-treat principle without adjusting for covariates. In secondary analyses, changes in ambulatory and clinical BP will be adjusted to assess the BP-independent effect of dietary sodium reduction on each subclinical CVD endpoint. The proposed trial has 85% statistical power to detect a clinically significant difference in changes of the four co-primary outcomes (10 g/m2 in LVMI, 1.3% in LVGLS, 0.9 m/s in cfPWV, and 1.1% in FMD) over 12 months between the two groups at a 2-sided significance level of 0.0125 (0.05/4). Findings from this trial will fill the knowledge gap of the underlying mechanisms of dietary sodium intake on CVD risk and provide further evidence on sodium reduction for CVD prevention.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥40 years. Individuals <40 years are at a low risk for clinical and subclinical CVD
* Elevated BP or hypertension (systolic BP ≥120 mmHg and diastolic BP ≥80 mmHg with or without use of antihypertensive medications)

Exclusion Criteria:

* Glomerular filtration rate (eGFR) <30 or end-stage renal disease (kidney transplant or chronic dialysis)
* History of cardiovascular disease
* Shift worker or regularly work at night
* Cancer requiring chemotherapy or radiation treatment in the previous two years
* Current pregnancy or breastfeeding or plans to become pregnant during the study
* Consumption of ≥21 alcoholic drinks/week
* Current participation in another lifestyle intervention or drug trial
* Current residence or planned residence that makes it difficult to meet trial requirements
* Other concerns regarding ability to meet trial requirements (at the discretion of the study coordinator)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Global Longitudinal Strain (LVGLS) from baseline to 12 months | 12 months
  Cardiac magnetic resonance imaging will be used to determine LVGLS.
Change in Left Ventricular Mass Index (LVMI) from baseline to 12 months | 12 months
  Cardiac magnetic resonance imaging will be used to determine left ventricular mass (LVM). LVM will be indexed to body surface area.
Change in Pulse Wave Velocity (PWV) from baseline to 12 months | 12 months
  A carotid tonometer will be used to measure carotid-femoral PWV.
Change in Flow-Mediated Dilation (FMD) from baseline to 12 months | 12 months
  Endothelial-dependent FMD will be quantified using high resolution ultrasound.

SECONDARY OUTCOMES:
Left Ventricular Volumes | Baseline, 6 months, and 12 months
  Cardiac magnetic resonance imaging will be used to determine left ventricular volumes.
Left Atrial Maximum and Minimum Volume | Baseline, 6 months, and 12 months
  Cardiac magnetic resonance imaging will be used to determine left atrial maximum and minimum volumes.
Left Atrial Ejection Fraction | Baseline, 6 months, and 12 months
  Cardiac magnetic resonance imaging will be used to determine left atrial ejection fraction.
Left Atrial Global Strain | Baseline, 6 months, and 12 months
  Cardiac magnetic resonance imaging will be used to determine left atrial global strain.
Aortic Pulse Wave Velocity | Baseline, 6 months, and 12 months
  Cardiac magnetic resonance imaging will be used to determine aortic pulse wave velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine T Mills, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Office of Health Research, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. The study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). Data will be prepared by the study coordinating center and sent to the PO for review prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, we will offer, through our public access website, opportunities for outside investigators to collaborate with us using complete study data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data sets will be submitted to the NHLBI Program Official (PO) no later than 3 years after the end of the final patient follow-up or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: Upon request